CLINICAL TRIAL: NCT06346574
Title: Changing the Culture of Health: Creating and Testing an Evidence-based Wellness Program for Diverse Head Start Centers, ABCD Head Start Randomized Control Trial: Healthy Eating, Activity, Relaxation Trial (HEART) at Head Start Pilot.
Brief Title: HEART at Head Start Pilot (Healthy Eating, Activity, Relaxation Trial)
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); National Head Start Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY-0004282
Record Dates: First submitted 2024-03-14; First posted 2024-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Dietary Habits; Physical Inactivity; Sleep Hygiene
Keywords: Health and Wellness app; Head Start educators; Guided goal setting; Motivational Interviewing for behavior change; Workplace wellness; Dietary habits; Physical inactivity; Sleep hygiene; Early Childhood Educators
MeSH Terms: conditions — Feeding Behavior; Sedentary Behavior; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Study participants will be educators at Head Start centers where either the intervention is offered at the onset of the study (intervention group) or after six months (comparison condition).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Behavioral:
  1. Access to health and wellness App from baseline to nine months.
  2. Access to Guides from baseline to six months
  Interventions: Behavioral: Experimental
- Delayed Intervention (Active Comparator): Behavioral:
  1. No access to health and wellness App from baseline to six months
  2. Access to App and Guide from six to nine months
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — Participants will receive access to health and wellness app and guide

SUMMARY:
With funding from the United States Department of Agriculture (USDA), the Tufts University's Friedman School of Nutrition Science and Policy will be implementing a new, health and wellbeing program for Head Start educators at ABCD Head Start Centers in the greater Boston area.

The purpose of this study is to evaluate the combined impact of a health and wellness program and behavior change guides. The evaluation will focus on ABCD Head Start educators as the study population. Tufts University's Friedman School of Nutrition Science and Policy is responsible for implementing and evaluating this new intervention through surveys and analysis of administrative (health and wellness App) data.

A paper and pencil survey will be used to gather information on dietary, physical activity, and sleep behaviors. The surveys will also include a module on satisfaction with the health and wellness App and Guides. Survey data will be combined with the administrative data about App utilization.

DETAILED DESCRIPTION:
Health and Wellness Apps can reduce barriers and increase access to health information. Supplemental coaching and support to set goals and work towards them may increase the likelihood of achieving physical activity and nutrition goals. This model of access to an App with supplemental support can be applied to improve the health and wellness of Head Start educators.

Head Start is the largest federally funded early childhood education program which provides an array of services to families in an early childhood care setting. The impact of Head Start on school readiness and nutritional outcomes of families has been examined extensively. There is growing awareness of the importance of supporting Head Start educators with their own health and wellness needs. There is a large volume of research that supports the use of Health and Wellness Apps.

The USDA awarded Tufts University a grant to develop, test, and evaluate an innovative health and wellness program for Head Start educators. Tufts University selected ABCD Head Start, which includes 19 Centers and approximately 250 educators in the greater Boston area. The team at Tufts University is leading the implementation and evaluation of the intervention, in collaboration with the National Head Start Association (NHSA) with ABCD Head Start as a community partner.

HEART at Head Start aims to generate evidence to inform how an innovative program can support the health and wellbeing of Head Start educators at the intervention centers compared to those at delayed intervention centers. Study participants will be provided access to the health and wellness app, which can either be downloaded onto mobile phones or accessed via the web. Users will be able to use a variety of health and wellness resources, webinars, as specialized coaching through this app. Additionally, Tufts guides will work closely with study participants to facilitate individual goal setting and to support work towards these set goals.

Evaluation findings will inform stakeholders about the feasibility of using a Health and Wellness App in conjunction with a guide to support Head Start educators with their health and wellness goals.

ELIGIBILITY:
Inclusion Criteria:

1. Educator at ABCD Head Start Center in the Greater Boston area
2. Ability to speak, read, and write in English fluently
3. Ability to download and use the Health and Wellness App on their mobile phone or computer
4. Residing in the US at the time of enrollment
5. Able to attend the baseline health fair at a ABCD Head Start Center

Study participants will be educators at ABCD Head Start centers where either the Health and Wellness App is offered at the onset of the study (intervention) or six months after the onset of the study (delayed intervention.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Use of health and wellness App | 9-months
  App based tracker use data
Engagement with Guide | 9-months
  Number of guide sessions attended
Nutrition behaviors | 9 months
  Self-reported food intake
Physical activity behaviors | 9 months
  Self-reported physical activity
Sleep habits | 9 months
  Self-reported sleep habits

SECONDARY OUTCOMES:
BMI | 9 months
  BMI values calculated using measured height and weight
Cholesterol | 9 months
  Non-fasting blood cholesterol obtained through finger prick method
Triglycerides | 9 months
  Non-fasting blood triglyceride obtained through finger prick method
Blood pressure | 9 months
  Measured systolic and diastolic blood pressure
Blood glucose | 9 months
  Non-fasting blood glucose obtained through finger prick method

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No